CLINICAL TRIAL: NCT02240212
Title: Phase Ib Study of Afuresertib Combined With Paclitaxel in Pre-treated HER2-negative Advanced Gastric Cancer
Brief Title: Study of Afuresertib Combined With Paclitaxel in Gastric Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: 201050
Record Dates: First submitted 2014-09-11; First posted 2014-09-15 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Cancer
Keywords: second line treatment; oncology; AKT inhibitor; paclitaxel; HER2 (ErbB2) negative advanced gastric cancer; Afuresertib
MeSH Terms: conditions — Neoplasms | interventions — afuresertib; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part 1: Dose-escalation (weekly paclitaxel) (Experimental): The dose escalation will be started from Cohort A (afuresertib combined with weekly paclitaxel regimen at 80 mg/m^2 d1, 8,15, q4w). The starting dose in Cohort A will be 125 mg afuresertib QD to indentify MTD
  Interventions: Drug: Afuresertib; Drug: Paclitaxel
- Part 1: Dose-escalation (3 weeks Paclitaxel) (Experimental): Once its MTD is identified, and then the study will move to dosing Cohort B (afuresertib combined with 3 weekly paclitaxel regimen at 175 mg/m^2 d1, q3w. Cohort B (afuresertib combined with 3 weekly paclitaxel regimen at 175 mg/m^2 d1, q3w). The starting daily dose of Cohort B will be 25 mg less than the MTD dose from Cohort A for afuresertib. If it is tolerated, then the dose escalation schedule will be followed in Cohort B until the MTD in this Cohort is reached. If the starting dose is not tolerated, then dose de-escalation will be explored until the MTD in this Cohort is reached. Once two dimensions of the MTD are achieved, then the optimal regimen for paclitaxel and MTD for afuresertib combined with paclitaxel based on the toxicity profile will be identified
  Interventions: Drug: Afuresertib; Drug: Paclitaxel
- Part 2: Experimental Cohort (Experimental): The optimal regimen for paclitaxel and MTD for afuresertib combined with paclitaxel based on the toxicity profile will be administered
  Interventions: Drug: Afuresertib; Drug: Paclitaxel

INTERVENTIONS:
Drug: Afuresertib — The unit dose strength is 50mg/75mg tablet. Afuresertib will be taken orally once daily continuously during trail.
Drug: Paclitaxel — Paclitaxel sourced locally will be administered IV

SUMMARY:
This is a Phase Ib, open-label, dose-escalation study to determine the Maximal tolerated dose (MTD) and the recommended Phase 2 dose (RP2D) for the combination of afuresertib and paclitaxel in subjects with recurrent HER2-negative gastric cancer, and further assess safety and preliminary efficacy of combination at the RP2D. Afuresertib had showed synergistic activity when combined with paclitaxel in vitro and in vivo models of gastric cancer. Dose escalation will continue until the MTD is established. The dose schedule is once daily (QD) dosing for afuresertib and intravenous (IV) infusion for paclitaxel Dose escalation in Part 1 will follow the 3 + 3 cohort design. A sequential approach will be conducted to explore the optimal paclitaxel regimen (weekly or 3weekly schedule) when combined with afuresertib. The dose escalation will be started from Cohort A (afuresertib combined with weekly paclitaxel regimen at 80 milligram (mg)/meter (m)^2 day1, 8,15, every 4 weeks (q4w). The starting dose in Cohort A will be 125 mg afuresertib QD. Once its MTD is identified, and then the study will move to dosing Cohort B (afuresertib combined with 3 weekly paclitaxel regimen at 175 mg/m^2 day1, every 3 week (q3w). The starting daily dose of Cohort B will be 25 mg less than the MTD dose from Cohort A for afuresertib. If it is tolerated, then the dose escalation schedule will be followed in Cohort B until the MTD in this Cohort is reached. If the starting dose is not tolerated, then dose de-escalation will be explored until the MTD in this Cohort is reached. Once two dimensions of the MTD are achieved, then the optimal regimen for paclitaxel and MTD for afuresertib combined with paclitaxel based on the toxicity profile will be identified. The combination regimen at the RP2D selected following Part I will be further investigated in its efficacy and safety in the Part II Expansion Cohort. Once a combination dose regimen for Part 2 has been determined, at least 20 and up to 40 subjects will be enrolled at the dose regimen selected following Part I. Overall response rate (ORR) will be evaluated using a Green-Dahlberg design. The design consists with one interim analysis. If less than 3 responses are observed in the initial 20 subjects, enrollment will be terminated due to futility; otherwise, the study will continue to meet the planned sample size of 40 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Provided signed written informed consent
* Male or female >=18 years of age with a diagnosis of Performance Status score of 0 or 1 according to the Eastern Cooperative Oncology at the time of signing the informed consent
* Able to swallow and retain orally administered study treatment
* Women of childbearing potential must have a negative serum pregnancy test within 7 days prior to the first dose of study treatment and agree to use effective contraception during the study. Men with a female partner of childbearing potential must have either had a prior vasectomy or agree to use effective contraception (Condom [during non-vaginal intercourse with any partner - male or female] OR Double-barrier method: condom and occlusive cap (diaphragm or cervical/vault caps) plus spermicidal agent (foam/gel/film/cream/suppository) [during sexual intercourse with a female]. Abstinence, defined as sexual inactivity consistent with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
* Adequate organ system functions at screening as Hematologic system (Absolute neutrophil count >=1.5 x 10^9/Litre (L), Hemoglobin >=9.0 gram (g)/deci (d)L, Platelets >=100 x 10^9/microL without transfusion in the past 7 days, prothrombin time/ international normalized ratio (PT/INR) and partial thromboplastin time (PTT) <=1.5 x Upper limit of normal [ULN]), Hepatic system (Total bilirubin <=1.0x ULN, Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) <=2.5x ULN), Metabolic system (Fasting Serum Glucose < 126 milli (m)g/dL [7 millimol/L], Hemoglobin A1C<=8%) and Renal system (Serum creatinine <= ULN, 24-hour urine creatinine clearance >=60 mL/minute [min])
* Histologically confirmed from the stomach or gastroeosophageal (GE) junction cancer with documented HER2-negative (defined as immunohistochemistry (IHC) 0-1+ or IHC2+ with a negative fluorescent in situ hybridization (FISH) test assessed by local or designated central lab) in primary or metastatic tumor tissue.
* Metastatic or locally advanced, unresectable disease.
* Subjects must have received first-line platinum/fluoropyrimidine doublet regimen for advanced gastric cancer and now exhibit progressive disease (PD), and must have recovered from any treatment-related toxicity. Note: prior XELOX, XP, FOLFOX, or SP (S-1+cisplatin)) treatment could be eligible, but prior-taxane are ineligible. Note: if patient is refractory or disease progression within 6 months of adjuvant treatment, then his previous treatment would be considered as first line treatment rather than adjuvant treatment, and then this patient could be enrolled into this study if other inclusion/exclusion criterion meets.
* Subjects shall have at least one measurable disease (i.e., present with at least one measurable lesion) by RECIST version1.1

Exclusion Criteria:

* History of another malignancy. Exception: Subjects who have been disease-free for 3 years, or subjects with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible.
* Prior PI3K-AKT- mammalian target of rapamycin (mTOR) pathway targeted therapy will not be eligible. (Note: prior vaccine and immunotherapy is allowed but must end at least 8 weeks prior to study treatment).
* Unresolved toxicity (Grade <=1) from prior chemotherapy with the exception of alopecia or anemia (Hemoglobin >9 g/dL).
* Subjects with uncontrolled brain metastases or spinal cord compression.
* Current use of warfarin for therapeutic anticoagulation (Note: low molecular weight heparin is permitted).
* Presence of an active gastrointestinal disease (not including gastric cancer), or other condition known to interfere significantly with the absorption, distribution, metabolism, or excretion of drugs. Prior gastrectomy is allowed.
* History of myocardial infarction, acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting or bypass grafting within six months of Screening.
* Pregnant or lactating female.
* Any serious and/or unstable pre-existing medical, psychiatric disorder or other conditions that could interfere with subject's safety, obtaining informed consent or compliance to the study procedures.
* Any prohibited medication(s) as Co-administration of afuresertib and medications which are a sensitive substrate of CYP3A4, OATP1B1 and BCRP with a low therapeutic index will be prohibited. Coadministration of afuresertib and medications which are a sensitive substrate of CYP2C8 with a low therapeutic index will be used with caution.
* History of Type 1 diabetes
* Any major surgery within the last four weeks.
* QTcF interval >=470 milliseconds (msec)s.
* known immediate or delayed hypersensitivity reaction or idiosyncratic reaction to drugs similar or related to afuresertib and taxanes.
* Any contraindications (as identified by the investigator) to the doses of paclitaxel defined in the protocol.
* Any history of reduction in standard of care paclitaxel dose for peripheral neuropathy.
* Known Human Immunodeficiency Virus (HIV) infection or active hepatitis B or C. (Note: active Hepatitis B virus (HBV) infection is defined as ALT/AST is above or equal to normal range or HBV deoxyribonucleic acid (DNA) >=2×10^3-4 international unit (IU)/mL; active Hepatitis C virus (HCV) infection is defined as HCV ribonucleic acid (RNA)+ and ALT/AST is above normal range). Antiviral therapy should be initiated before study treatment, and maintain during study treatment in patients with inactive HBV infection. Prophylaxis against HBV reactivation is recommended in accordance with established guidelines: the Asian-Pacific census statement on HBV in 2012 and Taiwan health insurance guidance in 2013.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2017-02-07 (Actual); Study Completion 2017-02-07 (Actual)

PRIMARY OUTCOMES:
Number of subjects with any serious adverse event (SAE), non-serious adverse event (AE) in Phase I Dose Escalation phase | Day 1 to Day 21 after the last dose of study treatment (assessed up to 1 years)
  An AE is defined as any untoward medical occurrence in a subject or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect
Assessment of changes in clinical laboratory tests in Phase I Dose Escalation phase | Day 1 to Day 21 after the last dose of study treatment. (assessed up to 1 years)
  Clinical laboratory tests included hematology, clinical chemistry, urinalysis
Assessment of 12-lead electrocardiogram (ECG) findings in Phase I Dose Escalation phase | Screening and Day 22
  Heart rate, pulse rate (PR), QRS, QT, and Electrocardiogram QT interval corrected for heart rate using Fridericia's formula (QTcF intervals) will be recorded by measuring triplicate 12-lead ECGs, obtained in semi-recumbent or supine position after 5 minutes rest
Assessment of Echocardiograms (ECHOs) in Phase I Dose Escalation phase | Every 9 weeks (for 3 weekly paclitaxel regimen) and every 8 weeks (for weekly paclitaxel regimen) until day 21 after last dose of study treatment (assessed up to 1 years)
  The cardiac ejection fraction and cardiac valve morphology will be assessed by ECHOs. The evaluation of the echocardiographer should include an evaluation for left ventricular ejection fraction (LVEF)
Assessment of blood pressure (vital signs) in Phase I Dose Escalation | Screening to Day 21 after the last dose of study treatment (assessed up to 1 years)
  Vital signs will include measurement of systolic and diastolic blood pressure. Vital signs should be measured after resting for at least 5minutes in a semi-supine position
Assessment of preliminary clinical efficacy in Phase II dose expansion | Every 6 weeks for 3 weekly paclitaxel regimen or every 8 weeks for weekly paclitaxel regimen (assessed up to 1 years)
  Tumor response will be measured by Response Evaluation Criteria In Solid Tumors (RECIST 1.1), the ORR will be based on confirmed responses by investigator-based assessment for gastric cancer
Assessment of respiration rate (vital signs) in Phase I Dose Escalation | Screening to Day 21 after the last dose of study treatment (assessed up to 1 years)]
  Vital signs will include measurement of respiration rate. Vital signs should be measured after resting for at least 5minutes in a semi-supine position.
Assessment of PR (vital signs) in Phase I Dose Escalation | Screening to Day 21 after the last dose of study treatment (assessed up to 1 years)]
  Vital signs will include measurement of PR. Vital signs should be measured after resting for at least 5minutes in a semi-supine position.

SECONDARY OUTCOMES:
Composite of pharmacokinetics parameters of afuresertib and paclitaxel combination regimen in dose escalation cohort | Day 1 (pre-dose, 1 to 3 hour [h]), Day 22 (pre-dose, 1 to 3 h and 6-8 h) for 3 weekly dose Paclitaxel regimen
  Afuresertib pharmacokinetic parameters following single and repeat dose administration, including Area under the concentration-time curve (AUC), Maximum observed concentration (Cmax) and paclitaxel Pre-dose (trough) concentration at the end of the dosing interval (Ctrough), Cmax after repeat dose administration, time of occurrence of Cmax (tmax), and terminal phase half-life (t1/2)
Evaluation of the progression free survival (PFS) in expansion cohort | Day 1and the earliest date of disease progression or death due to any cause; up to 6 months
  PFS is defined as the interval between first dose and the earliest date of disease progression or death due to any cause by investigator assessment
Number of subjects with any SAE, AE in expansion cohort | Day 1 to Day 21 after the last dose of study treatment (assessed up to 1 years).
  An AE is defined as any untoward medical occurrence in a subject or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect
Assessment of changes in clinical laboratory tests in expansion cohort | Day 1 to Day 21 after the last dose of study treatment (assessed up to 1 years)
  Clinical laboratory tests included hematology, clinical chemistry, urinalysis
Assessment of 12-lead ECG findings in expansion cohort | Screening and Day 22
  Heart rate, PR, QRS, QT, and Electrocardiogram QT interval corrected for heart rate using QTcF intervals will be recorded by measuring triplicate 12-lead ECGs, obtained in semi-recumbent or supine position after 5 minutes rest
Assessment of ECHOs in expansion cohort | Every 9 weeks (for 3 weekly paclitaxel regimen) or every 8 weeks (for weekly paclitaxel regimen) to day 21 after last dose of study treatment (assessed up to 1 years)
  The cardiac ejection fraction and cardiac valve morphology will be assessed by ECHOs The evaluation of the echocardiographer should include an evaluation LVEF
Assessment of composite pharmacokinetics of afuresertib and paclitaxel in expansion cohort | Day 1 (pre-dose, 1 to 3 hour [h]), Day 22 (pre-dose, 1 to 3 h and 6-8 h) for 3 weekly dose Paclitaxel regimen Day 1 (pre-dose, 1 to 3 h), Day 15 (pre-dose, 1 to 3 h and 6-8 h) for weekly dose Paclitaxel regimen
  Afuresertib concentration following single and repeat dose administration and Paclitaxel Ctrough and Cmax after repeat dose administration

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Novartis Investigative Site, Seoul, South Korea
- Novartis Investigative Site, Taipei, Taiwan